CLINICAL TRIAL: NCT06958250
Title: A Novel Endoscopic Bite Block
Brief Title: Novel Endoscopic Bite Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 857779
Record Dates: First submitted 2025-03-24; First posted 2025-05-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gastric Disease
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Novel Bite Block (Experimental): Insertion of Novel Endoscopic Bite Block in the subject's mouth following the usual manner prior to endoscopic procedure.
  Interventions: Device: Novel Bite Block

INTERVENTIONS:
Device: Novel Bite Block — The endoscopist will utilize the Novel Endoscopic Bite Block for the duration of the upper endoscopy (single-use, disposable).

SUMMARY:
This feasibility study aims to assess the safety and effectiveness of the Novel Endoscopic Bite Block. The device will be utilized in subjects undergoing routine outpatient upper endoscopy. The investigator hypothesizes that its innovative design will reduce complications associated with bite block positioning, thereby improving procedural efficiency and patient safety.

ELIGIBILITY:
Inclusion Criteria

1. Provision of a signed and dated Informed Consent Form (ICF).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, ≥21 years of age.
4. Deemed appropriate for scheduled upper endoscopy by endoscopists and anesthesia staff.

Exclusion Criteria

1. Known allergic reactions to thermoplastic polyurethane (TPU), the component used in the manufacturing of the Flexible Endoscopic Bite Block.
2. Any medical condition that, in the opinion of the PI, makes the subject ineligible to participate in the clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful completion of upper endoscopy procedures with the Novel Endoscopic Bite Block accessory | Day of procedure
  Proportion of endoscopic procedures that are successfully completed
Absence of dental injury during the upper endoscopy | Day of procedure
  Number and type of dental injuries occurred during the upper endoscopy

SECONDARY OUTCOMES:
Endoscopist's satisfaction with lack of bite block movement | Day of procedure
  Proportion of endoscopic procedures assessed by the endoscopist as satisfactory

CONTACTS AND LOCATIONS:
Overall Officials: Anish Sheth, MD, AGAF, Study Director — Penn Medicine Princeton Health
Locations (1):
- Penn Medicine Princeton Health, Plainsboro, New Jersey, United States